CLINICAL TRIAL: NCT02938793
Title: A Phase II Study of Durvalumab (MEDI4736) (Anti-PD-L1 Antibody) in Combination With Tremelimumab (Anti-CTLA-4 Antibody) in Subjects With Advanced Rare Solid Tumors
Brief Title: Durvalumab in Combination With Tremelimumab in Subjects With Advanced Rare Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor enrollment likely due to expanded availability of immunotherapy for patients
Sponsor: Prisma Health-Upstate (Other)
Collaborators: AstraZeneca (Industry); MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-15-11633
Record Dates: First submitted 2016-10-10; First posted 2016-10-19 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Rare Disease
Keywords: cancer, malignancy
MeSH Terms: conditions — Neoplasms; Rare Diseases | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Durvalumab, 1500 mg Q4W (equivalent to 20 mg/kg Q4W) intravenously for 13 doses and Tremelimumab 300mg intravenously as a single dose on cycle 1 day 1 only.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — intravenous administration
  Other Names: MEDI4736
Drug: Tremelimumab — intravenous administration
  Other Names: CP-675,206

SUMMARY:
This is an investigator initiated single institution, open-label study to evaluate the antitumor activity, safety, and tolerability of durvalumab in combination with tremelimumab in subjects with select advanced rare solid tumors.

DETAILED DESCRIPTION:
This is an investigator initiated single institution, open-label study to evaluate the antitumor activity, safety, and tolerability of durvalumab in combination with tremelimumab in subjects with select advanced rare solid tumors. The dose-exploration phase, conducted across a range of tumor types, has been completed. The dose-expansion phase is ongoing and includes certain soft tissue sarcomas, neuroendocrine tumors and thymic carcinoma. Therefore, subjects diagnosed with any of those rare tumors are excluded from this trial. Given the safety and tolerability data in the previous and ongoing studies (Study D4190C00010 and D4190C00006), the selected dose for evaluation in all subjects enrolled in this trial is as follows:

Durvalumab, 1500 mg Q4W (equivalent to 20 mg/kg Q4W) intravenously for 13 doses and Tremelimumab 300 mg intravenously as a single dose on cycle 1 day 1 only. Weight-based dosing should be utilized for patients <30 kg: durvalumab 20 mg/kg and tremelimumab 1 mg/kg. Tremelimumab will be administered first and the infusion duration will be approximately 1 hour. The durvalumab infusion will start approximately 1 hour after the end of the tremelimumab infusion and the infusion will be administered over approximately 1 hour.

The project Surveillance of Rare Cancers in Europe (RARECARE) collected data on cancers from 89 population-based cancer registries in 21 European countries, making it possible to study the epidemiology of these cancers as a whole in a large and heterogeneous population. Working from this database and the literature, a RARECARE working group produced a new list of cancers and developed a new definition of rare cancers (incidence < 6/100,000/year). This definition and working list are adopted for this rare tumor immunotherapy study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a rare advanced solid malignancy meeting EORTC criteria.
* Subjects must have failed or been ineligible to receive standard treatment options if available.
* Subjects must be amenable to biopsy of a tumor site or have recent (< 2 years) archival material available.
* ECOG performance status of 0 to 2.
* Life expectancy > 3 months.
* Adequate normal organ and marrow function including: hemoglobin > 9.0 g/dl; ANC > 1500 per mm3; platelet count > 100,000 per mm3; bilirubin < 1.5 x ULN; ALT/AST < 2.5 x ULN unless liver metastases present in which case must be < 5 x ULN; creatinine clearance > 40 ml/min by Cockcroft-Gault or 24 hour urine collection

Exclusion Criteria:

* Previous treatment with durvalumab or tremelimumab.
* Prior treatment with any checkpoint inhibitor (including anti-CTLA-4, anti-PD-1 and anti-PD-L1).
* Rare malignancies under investigation in other studies including thymic carcinoma, certain sarcomas, and neuroendocrine tumors.
* Untreated central nervous system metastatic disease.
* Active or documented autoimmune disease within previous 2 years.
* Uncontrolled psoriasis.
* Prior chemotherapy within 28 days of the first dose of durvalumab or tremelimumab.
* Steroid exposure within 28 days of the first dose of durvalumab or tremelimumab with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Antitumor Activity | 24 months
  To evaluate the antitumor activity of durvalumab in combination with tremelimumab based on immune-related Response Evaluation Criteria
Incidence of Treatment-Emergent and Non Treatment-Emergent Adverse Events [Safety and Tolerability] | 24 months
  To assess the safety and tolerability of durvalumab in combination with tremelimumab

SECONDARY OUTCOMES:
Expression of programmed cell death protein 1 (PD-1) | 24 months
  To evaluate the pharmacodynamic activity of durvalumab in combination with tremelimumab in the tumor microenvironment

CONTACTS AND LOCATIONS:
Overall Officials: William J Edenfield, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Greenville Health System Cancer Institute, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
aggregate data only

REFERENCES:
- [Background] Edenfield WJ, Chung K, O'Rourke M, Cull E, Martin J, Bowers H, Smith W, Gluck WL. A Phase II Study of Durvalumab in Combination with Tremelimumab in Patients with Rare Cancers. Oncologist. 2021 Sep;26(9):e1499-e1507. doi: 10.1002/onco.13798. Epub 2021 May 8. PMID 33893692